CLINICAL TRIAL: NCT00003352
Title: A Phase II Study in Patients With Metastatic or Locally Advanced Breast Cancer to Evaluate the Worth of the Combination of Adriamycin (Doxorubicin), Taxotere (Docetaxel), and Cyclophosphamide (ATC)
Brief Title: Combination Chemotherapy in Treating Women With Stage IIIB or Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP BP-58; NSABP-BP-58
Record Dates: First submitted 1999-11-01; First posted 2003-06-27 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cyclophosphamide — 600 mg/m2, IV, every 3 weeks
Drug: Taxotere — 60 mg/m2, IV, every 3 weeks
  Other Names: docetaxel
Drug: Adriamycin — 60 mg/m2, IV, every 3 weeks
  Other Names: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of doxorubicin, cyclophosphamide, and docetaxel in treating women with stage IIIB or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall response rate to doxorubicin, docetaxel, and cyclophosphamide (ATC) in women with metastatic or locally advanced breast cancer. II. Determine survival, time to first response, time to progression, and duration of response in these patients. III. Evaluate the feasibility of administering ATC for at least 4 courses. IV. Evaluate the toxicity profile of ATC and its effect on cardiac function.

OUTLINE: Patients receive intravenous doxorubicin over 15 minutes on day 0, followed by intravenous cyclophosphamide over 30 minutes. An hour after the end of the doxorubicin infusion, intravenous docetaxel is administered over 1 hour. Patients receive courses every 21 days until disease progression or unacceptable toxic effects are observed. When the maximum dose of doxorubicin is reached, treatment continues with docetaxel and cyclophosphamide. Patients with locally advanced breast cancer receive chemotherapy for at least 2 courses after documented response. Patients are followed every 6 weeks.

PROJECTED ACCRUAL: Approximately 89 patients will be accrued to this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic (stage IV) or locally advanced (stage IIIB) adenocarcinoma of the breast. Bidimensionally measurable disease. No active central nervous system (CNS) metastases. Brain metastases must be controlled for at least 3 months and have other sites of measurable disease. No carcinomatous meningitis. No lymphangitic lung metastases as the only site of metastatic disease. Hormone receptor status: Any estrogen or progesterone receptor status.

PATIENT CHARACTERISTICS: Age: 18 and over. Sex: Female. Menopausal status: Not specified. Performance status: Eastern Cooperative Oncology Group (ECOG) score range 0-2. Life expectancy: At least 6 months. Hematopoietic: Absolute neutrophil count at least 2,000/mm3. Platelet count at least 100,000/mm3. Hepatic: serum glutamic oxaloacetic transaminase (SGOT) and/or serum glutamic pyruvic transaminase (SGPT) no greater than 2.5 times upper limit of normal (ULN). Alkaline phosphatase no greater than 5 times ULN. Bilirubin no greater than ULN. No SGOT and/or SGPT greater than 1.5 times ULN if concomitant with alkaline phosphatase greater than 2.5 times ULN. Renal: Calcium no greater than 1.2 times ULN. Creatinine no greater than 1.5 times ULN. Cardiovascular:left ventricular ejection fraction (LVEF) at least institutional lower limit of normal on multiple gated acquisition scan (MUGA) or echocardiogram. No myocardial infarction within 6 months. No angina pectoris requiring antianginal medication. No history of congestive heart failure. No cardiac arrhythmias requiring medication. No vascular disease with documented cardiac function compromise No uncontrolled hypertension (diastolic greater than 100 mm Hg). Other: Not pregnant or nursing. Fertile patients must use effective barrier contraception. No diabetics with fasting blood sugar greater than 200 mg/dL. No peripheral neuropathy greater than grade 1. No psychosis or addictive disorders. No known hypersensitivity to E. coli-derived drugs.

PRIOR CONCURRENT THERAPY: Chemotherapy: No prior chemotherapy for metastatic breast cancer or non-breast cancer. At least 12 months since nontaxane containing adjuvant chemotherapy for primary tumor (in patients with metastatic disease). Prior adjuvant chemotherapy with anthracycline containing regimens allowed (provided total doxorubicin dose did not exceed 240 mg/m2). Endocrine therapy: At least 4 weeks since adjuvant hormone or hormone therapy for metastatic disease (at least 2 weeks for rapidly progressive disease). No concurrent hormonal birth control. Radiotherapy: At least 4 weeks since prior radiotherapy. Prior breast radiotherapy following lumpectomy allowed. No radiotherapy to greater than 30% of bone marrow. No prior left chest wall radiotherapy with anthracycline containing adjuvant chemotherapy. Surgery: Not specified.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 1998-06; Primary Completion 2000-09 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Best over-all tumor response that occurs during 6 cycles of chemotherapy | 18 weeks

SECONDARY OUTCOMES:
Survival | 18 weeks
Time to first response | 18 weeks
Time to progression | 18 weeks
Duration of response | 18 weeks
Completion of at least four cycles of chemotherapy | 12 weeks
Toxicity profile | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (166):
- United States (152):
  - Baptist Medical Center - Birmingham, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - Scripps Clinic and Research Foundation - La Jolla, La Jolla, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Saint Mary Medical Center - Long Beach, Long Beach, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Naval Medical Center - Oakland, Oakland, California
  - Sutter Cancer Center, Sacramento, California
  - Veterans Affairs Satellite Clinic - Sacramento, Sacramento, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Ocala Oncology Center, Ocala, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Winship Cancer Center, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Illinois Masonic Medical Center, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Highland Park Hospital, Highland Park, Illinois
  - West Suburban Hospital Medical Center, Oak Park, Illinois
  - Rockford Clinic, Rockford, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Methodist Cancer Center - Indianapolis, Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Norton Healthcare System, Louisville, Kentucky
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Regional Cancer Therapy Center - Frederick, Frederick, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. Louis University School of Medicine, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Albany Regional Cancer Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Genesee Hospital - Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Jewish Hospital of Cincinnati, Inc., Cincinnati, Ohio
  - Meridia South Pointe Hospital, Cleveland, Ohio
  - Mount Sinai Medical Center - Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Network - Bethlehem, Bethlehem, Pennsylvania
  - Penn State Geisinger Medical Center, Danville, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Kent County Memorial Hospital - Rhode Island, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Medical Group of Texas, Dallas, Texas
  - Kelsey Seybold Clinic, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Virginia Oncology Associates, Newport News, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Veterans Affairs Medical Center - Salem, Salem, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (12):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Manitoba Cancer Treatment and Research Foundation, Winnipeg, Manitoba
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Pavillion de Quebec, Québec, Quebec
  - Hopital Laval, Ste-Foy, Quebec
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan

REFERENCES:
- [Result] Smith RE, Anderson SJ, Brown A, Scholnik AP, Desai AM, Kardinal CG, Lembersky BC, Mamounas EP. Phase II trial of doxorubicin/docetaxel/cyclophosphamide for locally advanced and metastatic breast cancer: results from NSABP trial BP-58. Clin Breast Cancer. 2002 Dec;3(5):333-40. doi: 10.3816/CBC.2002.n.036. PMID 12533263